CLINICAL TRIAL: NCT03600987
Title: Effect of Music on Reading Comprehension in Patients With Aphasia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Carilion Clinic (Other)
Responsible Party: Principal Investigator, Jacqueline Treichler, ClinScD, CCC-SLP; Speech-Language Pathologist, Carilion Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB #2408
Record Dates: First submitted 2018-07-17; First posted 2018-07-26 (Actual); Last update posted 2020-01-06 (Actual); Status verified 2020-01

CONDITIONS: Aphasia
Keywords: left middle cerebral artery; cerebrovascular accident (CVA); stroke
MeSH Terms: conditions — Aphasia; Stroke

STUDY DESIGN:
Intervention Model Description: Single-subject adapted alternating treatment design.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Music and reading lyrics (Experimental): A single-subject adapted alternating treatment design will be used to compare two music conditions, using music with sung lyrics simultaneously with silent reading of the lyrics, and priming with music and sung lyrics followed by reading of the lyrics, with a control condition using reading materials without music.
  Interventions: Behavioral: Simultaneous music and reading lyrics; Behavioral: Priming with music; Behavioral: Control

INTERVENTIONS:
Behavioral: Simultaneous music and reading lyrics — listening to music with singing of the lyrics simultaneously with reading the written lyrics.
Behavioral: Priming with music — priming by listening to music and singing of the lyrics followed by reading the written lyrics.
Behavioral: Control — control condition using reading materials without music.

SUMMARY:
The purpose of this investigation is to examine the evidence on emotion, language, and music, and propose a first step, in the form of a single-subject research design, to determine the most effective and efficient method for application to the rehabilitation of patients with aphasia. A single-subject adapted alternating treatment design will be used to compare two music conditions, using music with sung lyrics simultaneously with reading of the lyrics, and priming with music and sung lyrics followed by a reading of the lyrics, with a control condition using reading lyrics without music. Results are expected to provide evidence of independent versus shared processing of music and language at the phrase level applied to the behavior of human subjects with aphasia.

DETAILED DESCRIPTION:
Quality assurance plan that addresses data validation and registry procedures, including any plans for site monitoring and auditing.

Data checks to compare data entered into the registry against predefined rules for range or consistency with other data fields in the registry.

Data verification to assess the accuracy, completeness, or representativeness of data by comparing the data to external data sources (reliability) Data dictionary: detailed descriptions of each variable Standard Operating Procedures: patient recruitment, data collection, data management, data analysis, reporting for adverse events change management. Sample size: A minimum of four participants will be required to demonstrate replication of treatment effects. A maximum of ten participants will be requested to account for attrition.

Plan for missing data, data inconsistency,or out-of-range results. Statistical analysis plan describing the analytical principles and statistical techniques to be employed in order to address the primary and secondary objectives, as specified in the study protocol or plan.

ELIGIBILITY:
Inclusion Criteria:

Post-hospitalization;

* premorbid reading at the 8th grade level or higher based on the participant's/family's stated years of formal education;
* post-stroke aphasia/left middle cerebral artery (MCA) cerebral vascular accident (CVA) based on electronic medical record (EMR) and computed tomography (CT) and/or magnetic resonance imaging (MRI) imaging reports, or consult with the neurologist;
* intact left amygdala and left extrastriate cortex based on EMR and CT/MRI imaging reports, or consult with the neurologist;
* reliability in answering yes-no questions as determined by an 80% score on therapy tasks during regular speech therapy;
* capacity to provide informed consent concerning a study involving an intervention with music therapy determined by the physician who refers the patient.

Exclusion Criteria:

* Co-morbidities diagnosed and reported in the EMR or shown on CT scan or MRI including past history of stroke in other brain regions with residual symptoms, dementia, Parkinson disease, head injury, etc.;
* hemianopsia or other visual field defects affecting vision for reading, and in particular right homonymous hemi- or inferior quadrantanopsia;
* previous history of learning disabilities in reading/writing;
* significant psychiatric diagnosis;
* English as a Second Language or non-English language.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2017-10-18 (Actual); Primary Completion 2019-10-17 (Actual); Study Completion 2019-10-17 (Actual)

PRIMARY OUTCOMES:
Percent correct responses per day on phrase completion task. | through study completion, an average of 1 year.
  Differential response to the interventions (counted as the percent correct responses per day).
Number of sessions required to achieve mastery. | through study completion, an average of 1 year.
  Count number of sessions.
Retention of the reading material. | 3 weeks post-intervention.
  Number of items recalled.

SECONDARY OUTCOMES:
International Classification of Functioning, Disability, and Health (ICF) body Functions/Structures, Activities, and Participation. | through study completion, an average of 1 year.
  Pretest-posttest information on the ICF Body Functions/Structures, Activities, and Participation (Hurkmans et al., 2011).
Boston Diagnostic Aphasia Examination-Third Edition (BDAE-3) (Goodglass, Harold, & Barresi, Austin: PRO-Ed.). | through study completion, an average of 1 year.
  BDAE-3 pretest-posttest reading scores on subtests: Word Identification/Word-Picture Match and Lexical Decision; Homophone Matching; Derivational and Grammatical Morphology/Matching to spoken sample; Oral Reading/Basic oral word reading; Oral Reading of Sentences with Comprehension; and Reading Comprehension-Sentences and Paragraphs. Pretest will be completed prior to baseline and initiating intervention, and posttest with be completed immediately following completion of intervention to assess generalization to non-trained stimuli.

CONTACTS AND LOCATIONS:
Overall Officials: Jacqueline A. Treichler, Principal Investigator — Carilion Clinic
Locations (1):
- Carilion Franklin Memorial Hospital, Carilion Community Memorial Hospital Inpatient Rehab, Carilion Day Rehab, Rocky Mount, Virginia, United States

IPD SHARING:
Plan to Share IPD: No
Share results without sharing protected health information or participant identification.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-03-30): https://cdn.clinicaltrials.gov/large-docs/87/NCT03600987/Prot_SAP_001.pdf